CLINICAL TRIAL: NCT03680300
Title: The Effectiveness of Muscle Energy Technique and Friction Massage in Hamstring Tightness Amongst Young Athletes of Pakistan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Isra University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IIRS-IUISB/M.PhilSMMPT/001
Record Dates: First submitted 2018-09-07; First posted 2018-09-21 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Hamstring Tightness; Hamstring Injury Prevention
Keywords: agility run test; vertical jump test; 100 meter sprint; nordic lower test; ymca sit and reach box; active knee extension; passive knee extension; post isometric relaxation; post facilitation stretch; muscle energy technique; friction massage; sports medicine; physical therapy; young athlete; pakistan

STUDY DESIGN:
Intervention Model Description: 60 athletes with hamstring tightness divided into 3 group.they will be Allocated by using a manual lottery system
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Post Facilitating Stretch (Experimental): Each patient in group A will be given with hot pack along with Tens for 20 mins then the patient will receive post facilitation stretch only, for about one month on daily basis.
  Interventions: Other: Post Facilitation Stretch
- Post Isometric Relaxation (Experimental): Each patient in group B will receive hot pack along with Tens for 20 mins then the patients will receive post isometric relaxation alone for about one months on daily basis.
  Interventions: Other: Post Isometric Relaxation
- Frictional Massage (Experimental): Frictional massage will be given to 3rd group
  Interventions: Other: Friction Massage

INTERVENTIONS:
Other: Post Facilitation Stretch — The Post Facilitating Stretch technique is performed as follows:
  The hamstring muscle will be placed between a fully stretched and a fully relaxed state. The patient will be asked to contract the agonist using a maximum degree of effort for 5-10 seconds while the therapist resists the patients force. The patient will then be asked to relax and release the effort, whereas the therapist will apply the rapid stretch to a new barrier and will be held for 10 seconds. Then the patient will relaxes for approximately 20 seconds and the procedure will be repeated between three to five times and five times more. Instead of starting from a new barrier, the muscle will be placed between a fully stretched and a fully relaxed state before every repetition.
  Arms: Post Facilitating Stretch
Other: Post Isometric Relaxation — The Post Isometric Relaxation technique is performed as follows :
  The hamstring muscle will be taken to a length just short of pain, or to the point where resistance to movement is first noted. A submaximal (10-20%) contraction of the hypertonic muscle will be performed away from the barrier for between 5 and 10 seconds and the therapist applies resistance in the opposite direction. The patient should inhale during this effort. After the isometric contraction the patient will be asked to relax and exhale while doing so. Following this a gentle stretch will be applied to take up the slack till the new barrier. Starting from this new barrier, the procedure is repeated two or three times.
  Arms: Post Isometric Relaxation
Other: Friction Massage — Each patient in group C will receive hot pack along with Tens for 20 mins then the patients will receive frictional massage alone for about one months on daily basis. Friction massage on hamstrings will be given for 20 mins by thrive massager by a therapist.
  Arms: Frictional Massage

SUMMARY:
The ability of an individual to move smoothly depends on his flexibility, an attribute that enhances both safety and optimal physical activity. Hamstring tightness leads to hamstring injuries and hamstring injuries are the most common type of injury among athletes. These injuries are slow to recover, make high health expenditure and decrease the performance level of the athlete.

The hamstring is an example of the muscle group that has a tendency to get shorten Muscle tightness is caused by a decrease in the ability of the muscle to deform, resulting in a decrease in the range of motion at the joint on which it acts. Inability to achieve greater than 120° of knee extension with the hip at 90° of flexion is considered as hamstring tightness.

DETAILED DESCRIPTION:
it will be a Randomized Controlled Trial with 3 group. there will be 60 patients with hamstring tightness divided into 3 group. Allocating by using the manual lottery system. Non-probability Convenience Sampling technique will be utilized. the self-structured questionnaire will be used to analyse the athletic condition and performance.

Each patient in group A will be given with hot pack along with Tens for 20 mins then the patient will receive post facilitation stretch only, for about one months on daily basis.

Each patient in group B will receive hot pack along with Tens for 20 mins then the patients will receive post isometric relaxation alone for about one months on daily basis.

Each patient in group C will receive hot pack along with Tens for 20 mins then the patients will receive frictional massage alone for about one months on daily basis. Friction massage on hamstrings will be given for 20 mins by thrive massager by a therapist.

ELIGIBILITY:
Inclusion Criteria:

* Athletes with Hamstring tightness
* Both male and female will be included.
* Athletes ages from 18 to 25 years
* Patients having Straight Leg Raise less then110˚

Exclusion Criteria:

* Athletes having hamstring injuries
* Patients having Straight Leg Raise greater then 110 ˚
* Above 25 years of age
* Other orthopedic condition like Low Back Pain,
* Athlete with any deformity Knee Joint

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2018-10-15 (Actual); Study Completion 2018-12-15 (Actual)

PRIMARY OUTCOMES:
Agility run test | one month
  performance test
vertical jump test | one month
  performance test
nordic lower test | one month
  performance test
ymca sit and reach box | one month
  performance test
Goniometer | one month
  passive straight leg raise range of motion
Goniometer | one month
  acticve Straight leg raise range of motion
Goniometer | one month
  active knee extension range of motion
Goniometer | one month
  passive knee extension range of motion

CONTACTS AND LOCATIONS:
Locations (1):
- Dr Abdul haseeb Bhutta, Mansehra, Khyber Pakhtoonkhawa, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Background] Payla M, Gill M, Singal SK, Shah N. A Comparison of the Immediate and Lasting Effects between Passive Stretch and Muscle Energy Technique on Hamstring Muscle Extensibility. Indian Journal of Physiotherapy & Occupational Therapy. 2018 Jan 1;12(1).